CLINICAL TRIAL: NCT02332772
Title: Prospective Study of Colonoscopic Resection of Large Polyps and Flat Lesions
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: PA14-0866
Record Dates: First submitted 2015-01-02; First posted 2015-01-07 (Estimated); Last update posted 2019-05-13 (Actual); Status verified 2019-05

CONDITIONS: Colon Polyps
Keywords: Colon Polyps; Large polyps; Flat lesions; Endoscopy; Colonoscopic resection; Colonoscopy; Data review; Data collection
MeSH Terms: conditions — Colonic Polyps | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Data Collection Endoscopy of Colon Polyps: Data collected from endoscopy reports and electronic medical record system to complete a descriptive analysis of the 1) demographics, 2) colonoscopy resection procedure, and 3) outcome of resection - immediate and delayed complications, tumor recurrence, and cancer during follow-up 01/01/2014 - 12/31/2025.
  Interventions: Other: Data Collection

INTERVENTIONS:
Other: Data Collection — Data collected from endoscopy procedures.

SUMMARY:
With this study, the investigators plan to review the performance of colonoscopic resection of large (> 1 cm) and flat lesions in the colon. The findings will help us define the role of colonoscopic resection of colon polyps and flat lesions and identity areas for improvement. The data will be used for continuing quality improvement and presenting our outcomes at academic meetings and publishing our results in peer reviewed journals.

DETAILED DESCRIPTION:
Our goal is to collect data from our endoscopy reports (Endoscopy Clinic database) and electronic medical record system (Clinic Station) to complete a descriptive analysis of the 1) demographics, 2) colonoscopy resection procedure, and 3) outcome of resection - immediate and delayed complications, tumor recurrence, and cancer during follow-up 01/01/2014 - 12/31/2025.

Specific variable to be reviewed:

1. Patient Demographics: Age, Sex, Race, Height, Weight, BMI (patient privacy will be acknowledged).
2. Indications for Colonoscopy (screening, surveillance, symptoms or tertiary referral [EMR])
3. Comorbid conditions: cancer and surgical history, medical conditions.
4. Colonoscopy procedure: Quality of colon preparation (using the Boston Bowel Preparation Scale) 0 - 3 for each section of the colon (Ascending, Transverse, Descending and Total Colon), cecal intubation rate, cecal intubation and total procedure time, type of colonoscope (if CO2 was used in the procedure and techniques for colonoscope insertion, including position changes.
5. Examination findings: Number of polyps and nature of polyps removed (site, size, surface, vascular pattern); type of polyp removed (serrated and sessile (flat); optical features and histology of polyps.
6. Resection techniques: Biopsy, snare resection, endoscopic mucosal resection, endoscopic submucosal dissection etc.
7. Including Pathology report findings so that a comparison can be made of the optical features and actual pathology report.
8. Outcomes of colonoscopy: Complete or incomplete resection, local recurrence, need for surgery, etc
9. Outcome of colonoscopy: Complications (Bleeding and perforation).

ELIGIBILITY:
Inclusion Criteria:

1. All Patients who have been referred for endoscopic resection of large polyps (>1 cm) and flat lesions.

Exclusion Criteria:

N/A

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing endoscopy at MD Anderson Cancer Center in Houston, Texas
Sampling Method: Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2015-04 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Composite Data Review of Colonoscopic Resection of Colon Polyps and Flat Lesions | 1 day
  Descriptive tables presented for demographics, polyp counts, colonoscopy experiences, polyp removals and findings. Proportions presented with 95% confidence intervals.
  Continuous values such as age and times presented with median, minimum and maximum.
  Comparisons among patient subgroups made with chi-square tests for categorical data and t-tests or the non-parametric alternative, Wilcoxon tests, to compare continuous measures.
  Graphics such as box plots, trellis plots, bar graphs, or stacked bar graphs used to describe distributions overall and among subgroups.

CONTACTS AND LOCATIONS:
Overall Officials: Gottumukkala S. Raju, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org